CLINICAL TRIAL: NCT06572943
Title: The Effect of Long-Term Moderate Intensity Exercise During Pregnancy on Maternal and Fetal Cardiovascular System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: George Makrydimas (Other)
Responsible Party: Sponsor-Investigator, George Makrydimas, Professor of Obstetrics and Gynaecology, University Hospital, Ioannina
Organization: University Hospital, Ioannina (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 3/30-01-2024 (θ. 6)
Record Dates: First submitted 2024-08-20; First posted 2024-08-27 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Pregnancy Related
Keywords: pregnancy; physical activity; exercise; Maternal cardiovascular system; Fetal cardiovascular system
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Routine Antenatal Care. Brochures with dietary recommendations will be given.
- Experimental (Experimental): Detailed recommendations and brochures regarding physical activity will be given.Moreover brochures with dietary recommendations will be administrated.
  Interventions: Other: Moderate intensity physical activity

INTERVENTIONS:
Other: Moderate intensity physical activity — Moderate intensity exercise of 30 minutes for at least 4-5 times per week (if not daily).
  Arms: Experimental

SUMMARY:
The investigators aim to evaluate the effect of long-term moderate intensity physical activity during pregnancy in maternal and fetal cardiovascular system. A randomized clinical trial was designed with two groups (Study group and Control Group).

DETAILED DESCRIPTION:
Physical activity (PA) enhances not only physical but also mental health.PA contributes to the prevention of a variety of diseases in general population including hypertension, diabetes mellitus, stress, and depression. Nevertheless, pregnancy is a time period that various changes take place in a woman's body. Those alterations might be either facilitators or barriers for conducting PA during pregnancy.

When it comes to pregnancy several benefits have been associated with PA for both mother and fetus; such as low gestational weight gain, lower incidence of gestational diabetes mellitus (GDM), better management of Pre-eclampsia and post-partum weight retention. Moreover, PA improves mental health in pregnant women, while recent studies have revealed that physical exercise during pregnancy can improve oxidative stress, inflammation and endothelial function. The vast majority of Obstetricians & Gynecologists recommend that pregnant women should be urged to start or continue doing physical activity in the absence of contraindications. To be more specific, pregnant women should do at least 150 minutes of moderate intensity PA weekly. However, several studies support that pregnant women all over the world does not meet those recommendations. Relevant evidence of published literature are scarce regarding the alterations on maternal and fetal cardiovascular system due to chronic exercise .

Thus, investigators aim to evaluate the effect of long-term moderate intensity PA in maternal and fetal cardiovascular system. Thus, a randomized clinical trial with two groups (study group-control group) was designed. The study group includes pregnant women during the 1st trimester that will undergo moderate intensity PA, while the control group includes pregnant women that will receive the routine antenatal care. Participants will be followed up until 6 months postpartum.

To be more specific, all participants will receive a pedometer to record their daily steps from the first trimester until the postpartum period. The intervention group will additional receive detailed recommendations for 30 minutes of moderate intensity exercise at least 4-5 times per week (if not daily) and brochures with relevant information will be administrated as well. Moreover, brochures with dietary recommendations during pregnancy will be given to all participants.

Three routine antenatal ultrasound scans at 11-13+6 , 20-24, and 32-36 gestational weeks will be performed. Maternal Uterine Dopplers will be assessed at every scan, while fetal Dopplers will be done at 2nd and 3rd trimester. Maternal cardiovascular assessment will take place at 1st trimester, 3rd trimester and postpartum with transthoracic echocardiography, ophthalmic artery Doppler, Flow Mediated Dilatation and Arterial Stiffness . Fetal heart function will be assessed at 2nd and 3rd trimester. Evaluation of the infants' heart will also be performed at 6 months postpartum. A questionnaire evaluating mental health known as Depression-Anxiety and Stress Scale 21 (DASS-21) in pregnant women will be administered during the 1st and 3rd trimester. Maternal body fat measurements will take place at each trimester and postpartum. In addition fat composition of both the fetus will be evaluated by ultrasound before the delivery and the newborn within 48 hours following birth. Maternal blood sample will be collected during 1st trimester, 3rd trimester and postpartum and blood sample from the umbilical cord during labour, to assess several parameters.

All participants will be fully informed about the purpose of the study and will be included only after signing the Informed Consent Form. All data collected will be confidential and only accessible to members of the research team. These data will be coded according to GDPR. The clinical implementation of this study will be according to the International Code of Medical Ethics of the World Medical Association (Declaration of Helsinki), and all participants submitted a written informed consent since a detailed description of all aspects and the objectives of the study are explained and fully understood. The ethical committee of the University Hospital of Ioannina approved this study (decision number: 3/30-01-2024; date of approval; 30 January 2024).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women during 1st trimester, who had the routine dating scan at 11-13+6 gestational weeks [also known as Nuchal translucency (NT) scan] and the uterine arteries (UtA) PI assessment

Exclusion Criteria:

* Diabetes Mellitus (Type I or II)
* Maternal age < 18 years old
* Body Mass Index (BMI) > 40
* Contraindications for PA: Multiple Pregnancies, Vaginal Bleeding, Hypertension or Gestational Hypertension, Uncontrolled Thyroid Diseases, Cardiovascular Diseases (e.g. valvular diseases, congenital heart diseases, cardiomyopathies, atrial fibrillation, coronary heart disease) or respiratory system diseases (asthma, chronic obstructive pulmonary disease) or systemic disease (cancer, autoimmune diseases) or several other diseases considered to be barriers for PA during pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-26 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Uterine Arteries Pulsatility Index at each trimester | 11-13+6, 20-24, and 32-36 gestational weeks
  Uterine Arteries Pulsatility Index will be measured with Ultrasound Doppler by the same operator, at each trimester

SECONDARY OUTCOMES:
Umbilical artery Pulsatility Index during the 2nd and 3rd trimester | 20-24, and 32-36 gestational weeks
  Measured with Ultrasound Doppler by the same operator
Middle Cerebral Artery Pulsatility Index during the 2nd and 3rd trimester | 20-24, and 32-36 gestational weeks
  Measured with Ultrasound Doppler by the same operator
Incidence of Gestational Diabetes | 26-29 weeks gestation
  Diagnosis will be made based on oral glucose tolerance test with ingestion of 75g of glucose. Abnormal is considered either of the following: fasting glucose >92mg/dl, glucose >180mg/dl one hour after, glucose >153mg/dL two hours after.
Incidence Pre-eclampsia | >20 weeks until 4-6 weeks postpartum
  New onset of hypertension and proteinuria or the new onset of hypertension plus significant end-organ dysfunction with or without proteinuria
Maternal body fat measurements | 11-13+6., 20-24, and 32-36 gestational weeks, 8-12 weeks postpartum
  Measured with calibrated body fat scale
Gestational weight Change | Between 36-40 weeks gestation
  Comparison of maternal weight at the time of inclusion in the study and at the final ultrasound examination.
Gestational age at labor | Delivery
  Gestational weeks
Maternal mental health | 11-13+6. and 32-36 gestational weeks
  Depression-Anxiety and Stress Scale 21. This scale is a 21 item self report questionnaire designed to measure the severity of a range of symptoms common ot both Depression and Anxiety. Each item is scored from 0 (did not apply to me) to 3(applied to me very much or most of the time). The scale ot which each item belongs is indicated by the letters D(Depression), A(Anxiety) and S (Stress). For each scale (D, A&S) sum the scores for identified items. The higher scores indicate more severe conditions.
Maternal cardiovascular adaptations during pregnancy and postpartum | 11-13+6, 32-36 gestational weeks and 8-12 weeks postpartum
  Transthoracic echocardiography will be performed by specialist cardiologist and will assess the following parameters: PWV, cSBP, cPP, LVEF, LVEDd, LVM, GLS, EDV, ESV, LAV, LAVI, MPI, LVMI, IVS, VTI, TR, PWT, RWT, E wave velοcity, A wave velocity, Deceleration time E/A ratio, Lateral e' velocity, Septal e' velocity
Arterial stiffness and FMD adaptations thorough pregnancy | 11-13+6. and 32-36 gestational weeks and 8-12 weeks postpartum
  : Arterial Stiffness will be evaluated using the Mobil-O-Graph tool as assessed by the Pulse wave Velocity (PWV). FMD represents a non-invasive method to determine the endothelial dysfunction in the brachial artery in response to reactive hyperaemia.
Maternal Blood Samples' findings | 11-13+6, 32-36 gestational weeks and 8-12 weeks postpartum
  : Maternal blood samples will be analyzed by certified laboratories and the findings will be evaluated. Comparisons between the two groups will take place.
Umbilical cord blood samples; findings | Delivery
  Umbilical cord blood samples will be analyzed by certified laboratories and the findings will be evaluated. Comparisons between the two groups will take place
Fetus and Neonatal Fat Composition | Before delivery and within 48 hours following delivery
  Fat composition of the neonate will be measured with ultrasound at the level of femur, humerus abdomen and scapula. Comparisons between the two groups will take place
Fetal heart adaptations and cardiovascular changes of the infant | 20-24, 32-36 gestational weeks and 5-7 months postpartum.
  The following parameters were obtained via fetal echocardiography during ultrasound examinations at 20-24 and 32-36 gestational weeks as well as transthoracic echocardiography of the infant at 5-7 months old: MAPSE, TAPSE, LVCO, LVEF, E/A ratio, AoI PI, DA PI, Aorta peak velocity, Pulmonary Artery peak Velocity. A comparison between the two groups (study group-control group) will be conducted, as well.

CONTACTS AND LOCATIONS:
Overall Officials: George Makrydimas, Professor, Study Director — University Hospital, Ioannina
Locations (1):
- Department of Obstetrics and Gynecology, University Hospital of Ioannina, Ioannina, Greece

REFERENCES:
- [Background] Martland R, Mondelli V, Gaughran F, Stubbs B. Can high-intensity interval training improve physical and mental health outcomes? A meta-review of 33 systematic reviews across the lifespan. J Sports Sci. 2020 Feb;38(4):430-469. doi: 10.1080/02640414.2019.1706829. Epub 2019 Dec 31. PMID 31889469
- [Background] Zschucke E, Gaudlitz K, Strohle A. Exercise and physical activity in mental disorders: clinical and experimental evidence. J Prev Med Public Health. 2013 Jan;46 Suppl 1(Suppl 1):S12-21. doi: 10.3961/jpmph.2013.46.S.S12. Epub 2013 Jan 30. PMID 23412549
- [Background] Davies G, Artal R. It's time to treat exercise in pregnancy as therapy. Br J Sports Med. 2019 Jan;53(2):81. doi: 10.1136/bjsports-2018-100360. Epub 2018 Dec 15. No abstract available. PMID 30554145
- [Background] Michalek IM, Comte C, Desseauve D. Impact of maternal physical activity during an uncomplicated pregnancy on fetal and neonatal well-being parameters: a systematic review of the literature. Eur J Obstet Gynecol Reprod Biol. 2020 Sep;252:265-272. doi: 10.1016/j.ejogrb.2020.06.061. Epub 2020 Jun 29. PMID 32634674
- [Background] Physical Activity and Exercise During Pregnancy and the Postpartum Period: ACOG Committee Opinion, Number 804. Obstet Gynecol. 2020 Apr;135(4):e178-e188. doi: 10.1097/AOG.0000000000003772. PMID 32217980
- [Background] Mottola MF, Davenport MH, Ruchat SM, Davies GA, Poitras VJ, Gray CE, Jaramillo Garcia A, Barrowman N, Adamo KB, Duggan M, Barakat R, Chilibeck P, Fleming K, Forte M, Korolnek J, Nagpal T, Slater LG, Stirling D, Zehr L. 2019 Canadian guideline for physical activity throughout pregnancy. Br J Sports Med. 2018 Nov;52(21):1339-1346. doi: 10.1136/bjsports-2018-100056. PMID 30337460
- [Background] Evenson KR, Wen F. Prevalence and correlates of objectively measured physical activity and sedentary behavior among US pregnant women. Prev Med. 2011 Jul-Aug;53(1-2):39-43. doi: 10.1016/j.ypmed.2011.04.014. Epub 2011 May 4. PMID 21575654
- [Background] Hesketh KR, Evenson KR. Prevalence of U.S. Pregnant Women Meeting 2015 ACOG Physical Activity Guidelines. Am J Prev Med. 2016 Sep;51(3):e87-9. doi: 10.1016/j.amepre.2016.05.023. No abstract available. PMID 27544437
- [Background] Fernandez-Buhigas I, Martin Arias A, Vargas-Terrones M, Brik M, Rolle V, Barakat R, Munoz-Gonzalez MD, Refoyo I, Gil MM, Santacruz B. Fetal and maternal Doppler adaptation to maternal exercise during pregnancy: a randomized controlled trial. J Matern Fetal Neonatal Med. 2023 Dec;36(1):2183759. doi: 10.1080/14767058.2023.2183759. PMID 36889747
- [Background] Chatzakis C, Sotiriadis A, Fatouros IG, Jamurtas AZ, Deli CK, Papagianni M, Dinas K, Mastorakos G. The Effect of Physical Exercise on Oxidation Capacity and Utero-Placental Circulation in Pregnancies with Gestational Diabetes Mellitus and Uncomplicated Pregnancies, a Pilot Study. Diagnostics (Basel). 2022 Jul 16;12(7):1732. doi: 10.3390/diagnostics12071732. PMID 35885635
- See also: Exercise Holds Even More Heart Health Benefits for People with Stress-Related Conditions. American College of Cardiology — https://www.acc.org/About-ACC/Press-Releases/2022/03/23/18/18/http%3a%2f%2fwww.acc.org%2fAbout-ACC%2fPress-Releases%2f2022%2f03%2f23%2f18%2f18%2fExercise-Holds-Even-More-Heart-Health-Benefits-for-People-with-Stress-Related-Conditions.
- See also: Exercise in Pregnancy — https://linkinghub.elsevier.com/retrieve/pii/S0278591917300522
- See also: Physical activity and pregnancy. RCOG — https://www.rcog.org.uk/for-the-public/browse-all-patient-information-leaflets/physical-activity-and-pregnancy/